CLINICAL TRIAL: NCT04181775
Title: Effectiveness of an ADE-related Hospitalization Risk Prediction Tool for Patients Discharged from the Emergency Department (ADE-RED)
Brief Title: Effectiveness of an ADE-related Hospitalization Risk Prediction Tool for Patients (ADE-RED)
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 060.PHA.2019.A
Record Dates: First submitted 2019-11-27; First posted 2019-11-29 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Adverse Drug Event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: ADE-RED scoring tool — The ADE-RED scoring tool will reduce the incidence of future visits to the ED or future admissions by identifying patients who are at high risk for ADE-related readmissions.

SUMMARY:
The rationale for this study is to evaluate the effectiveness of a risk prediction tool for patients who are at high risk for ADEs resulting in hospitalization or ED revisit. The ADE-RED score initiates a PLMR that literature has shown reduces medication discrepancies and ADEs at hospital admission and discharge. No current system identifies patients presenting to the ED that may benefit from PMLR independent of an admission disposition. The ADE-RED scoring tool will reduce the incidence of future visits to the ED or future admissions by identifying patients who are at high risk for ADE-related readmissions.

DETAILED DESCRIPTION:
There has been considerable attention placed on adverse drug events (ADEs) and their effects on readmission rates worldwide. Several studies have tried to identify the drugs most commonly responsible for ADEs, high-risk patient populations, and the causes of these ADEs. Some of the causes that have been postulated include the aging population, increasing number of drugs on the market, and a troubling upward trend in polypharmacy. The reported rates of ADE-related hospitalizations have varied from study to study. Kongkaew et al. estimated around 5% of all hospital admissions are the result of an adverse drug reaction (ADR), which is a subtype of ADEs. Meanwhile, Shehab et al. estimated approximately 27.3% of emergency department (ED) visits for ADEs result in hospitalization.

Unfortunately, practitioners may exacerbate the problem by prescribing additional pharmacotherapy for conditions caused by an unrecognized ADE. Such circumstances can lead to additional cost and harm to patients. However, pharmacists are uniquely qualified to recognize and address potential ADEs through pharmacist-led medication reconciliation (PLMR). PLMR is the process in which a pharmacist produces an accurate list of medications a patient is taking and compares that list against the patient's documented admission, transfer, and/or discharge orders. Several years of education and training to learn the pharmacokinetic and pharmacokinetic characteristics of a wide variety of medications, as well as any potential side effects, have given pharmacists the skills to detect, assess, and understand ADEs. Many institutions have implemented PLMRs within specific hospital units, such as the ED, in an effort to increase cost savings to the patient and the health care institution.

A meta-analysis of patients with preventable ADEs found that as much as 52% of ADEs, present at the time of hospitalization or an emergency visit, were preventable (8). This highlights the need to produce a tool to predict patients at risk for ADE-related hospitalizations. There have been several ADE risk prediction initiatives developed to identify high risk patients (9-17). Many of these risk prediction tools, such as the Prediction of Hospitalization due to ADRs in Elderly Community-Dwelling Patients (PADR-EC) score and the Brighton Adverse Drug Reactions Risk (BADRI) model, focused on older patients, hospitalized patients, or both. A focus on prediction tools in older adults is reasonable due to ADE-related hospitalization rates among adults 65 years or older, being seven times higher than adults younger than 65 years old (6). However, there is limited information in risk scoring tools for the general public who present to the ED and are at high risk of an ADE. In 2017, a Transitions of Care pharmacy resident at Methodist Dallas Medical Center (MDMC) developed a risk scoring tool to help identify patients in the ED who were at high risk for an ADE-related hospitalization. The scoring tool, which was named the ADE-RED score, took into account the patient's age, presence of polypharmacy, specific high- risk medications, number of previous ED visits, comorbidities, and the reason for their current visit. A score of 12 or more alerted ED pharmacists to perform a PLMR and to make necessary interventions and recommendations to medical staff. Therefore the ADE-RED program has the opportunity to fill a gap in the care for patients who may be hospitalized or return to the ED due to a preventable ADE.

This study will be conducted to determine whether the ADE-RED score can reduce the incidence of ADE- related readmissions compared to the incidence of such readmissions as observed from sister facilities within the Methodist Health System (MHS) and to determine whether the ADE-RED score can predict patients at risk of readmission.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hospital with a prior ED visit within the previous 30 days
* Patients presenting to the ED with a prior ED visit within the previous 30 days

Exclusion Criteria:

* Patients without PTA medications at the time of initial ED presentation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are considered high risk if the score is > 12, moderate risk if the score 6-11, and low risk if the score is 0-5. High-risk patients are flagged in the electronic medical record of the patient, alerting the pharmacist to complete a medication reconciliation and address any issues.
Sampling Method: Non-Probability Sample
Enrollment: 471 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Incidences of ADE-related readmission within 30 days of prior ED visit. | one month period in March 2019
  Incidences of ADE-related readmission within 30 days of prior ED visit.

SECONDARY OUTCOMES:
Percentage of patients who were readmitted who did or did not have an ADE-RED score at initial ED visit. | one month period in March 2019
  Percentage of patients who were readmitted who did or did not have an ADE-RED score at initial ED visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ilka Ratsaphangthong, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided